CLINICAL TRIAL: NCT02130362
Title: A Long-Term Non-Interventional Postmarketing Study to Assess Safety and Effectiveness of Humira® (Adalimumab) in Pediatric Patients With Moderately to Severely Active Crohn's Disease (CD) - CAPE
Brief Title: A Non-Interventional Clinical Study to Evaluate Long-Term Safety and Effectiveness of HUMIRA (Adalimumab) in Pediatric Patients With Moderately to Severely Active Crohn's Disease (CD)
Acronym: CAPE
Status: Active, not recruiting | Type: Observational
Sponsor: AbbVie (Industry)
Responsible Party: Sponsor
Other Study IDs: P11-292
Record Dates: First submitted 2014-05-01; First posted 2014-05-05 (Estimated); Last update posted 2025-07-16 (Actual); Status verified 2025-07

CONDITIONS: Crohn's Disease
Keywords: Crohn's Disease; Registry; Adalimumab; Crohn's; Inflammatory Bowel Diseases; Gastrointestinal Diseases
MeSH Terms: conditions — Crohn Disease; Inflammatory Bowel Diseases; Gastrointestinal Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Immunosuppressant Therapy: Pediatric patients who are being prescribed and treated with immunosuppressant therapy
- Adalimumab (Humira) Treatment: Pediatric patients who are prescribed and treated with adalimumab

SUMMARY:
This is a registry study to evaluate the long-term safety and effectiveness of adalimumab in pediatric patients with moderately to severely active CD who are treated as recommended in the local product label.

ELIGIBILITY:
Inclusion Criteria:

* For a patient enrolling into the HUMIRA treatment group; A pediatric patient between the ages of 6 and 17 years inclusive at the time of enrollment, diagnosed with moderately to severely active CD who has been prescribed Humira therapy according to the routine clinical practice.
* For a patient enrolling into the immunosuppressant therapy treatment group; A pediatric patient between the ages of 6 and 17 years inclusive at the time of enrollment, diagnosed with moderately to severely active CD who has been prescribed azathioprine, 6-mercaptopurine or methotrexate.
* Parent or guardian; or patient (if 18 years of age or older at enrollment and rolling over from an AbbVie-sponsored investigational Pediatric CD investigation trial) has voluntarily signed and dated an Authorization for Use/Disclosure of Data (AUDD)/informed consent form (ICF) after the nature of the registry has been explained and the patient, patient's parent or legal guardian has had the opportunity to ask questions.

Exclusion Criteria:

* Patients should not be enrolled into the registry if they are currently being treated with any investigational agents or are receiving any investigational procedures.
* Patients should not be enrolled into the immunosuppressant therapy treatment group if they require ongoing treatment with approved biologic agents including HUMIRA.

Ages: 6 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Pediatric patients with moderately to severely active Crohn's Disease (CD) who have been prescribed HUMIRA according to the local label and pediatric patients being prescribed and treated with IMM (azathioprine, 6-mercaptopurine, or methotrexate). Patients being prescribed and treated with immunosuppressant therapy with no concurrent biologic use will be enrolled as a reference group.
Sampling Method: Probability Sample
Enrollment: 1446 (Actual)
Dates: Start 2014-08-28 (Actual); Primary Completion 2030-11 (Estimated); Study Completion 2030-11 (Estimated)

PRIMARY OUTCOMES:
Number of treatment-emergent AESI per 100 PYs of infections and malignancies | Up to 10 years
Percentage of subjects with SAEs | Up to 10 years
Number of treatment-emergent other AESI per 100 PYs | Up to 5 years
Percentage of subjects with other AESI | Up to 5 years
  Percentages of subjects with AESIs other than infections and malignancies
Number of subjects with Adverse Events of Special Interest (AESI) of infections, malignancies, and pregnancies | Up to 10 years
Number of subjects with other AESI | Up to 5 years
  Number of subjects with AESIs other than infections and malignancies
Number of treatment-emergent SAEs per 100 patient years (PYs) | Up to 10 years
Number of subjects with Serious Adverse Events (SAEs) | Up to 10 years
Percentage of subjects with AESI of infections, malignancies, and pregnancies | Up to 10 years

SECONDARY OUTCOMES:
Short Pediatric Crohn's Disease Activity Index (sh-PCDAI) | Up to 5 years
  Patient completed questionnaires
Short Quality of Life in Inflammatory Bowel Disease Questionnaire (SIBDQ) | Up to 5 years
  Completed by the patients who are 18 years of age or older
Work Productivity and Activity Impairment (WPAI) questionnaire | Up to 5 years
  Completed by caregiver up to the age of 17 years and completed by the patients of age 18 years or above.
Physician's Global Assessment of Disease Activity (PGA) | Up to 5 years
  Completed by the physician
IMPACT III | Up to 5 years
  Completed by patients ages 10 through 17 years old

CONTACTS AND LOCATIONS:
Overall Officials: ABBVIE INC., Study Director — AbbVie
Locations (148):
- United States (45):
  - Univ Alabama, Birmingham CCC /ID# 146060, Birmingham, Alabama
  - University of South Alabama /ID# 137255, Mobile, Alabama
  - Phoenix Children's Hospital /ID# 141336, Phoenix, Arizona
  - Children's Hospital Los Angeles /ID# 141551, Los Angeles, California
  - Private practice: Dr. Shervin Rabizadeh /ID# 137269, Los Angeles, California
  - Rady Children's Hospital San Diego /ID# 140883, San Diego, California
  - Univ California, San Francisco /ID# 141312, San Francisco, California
  - Children's Hospital Colorado - Aurora /ID# 137261, Aurora, Colorado
  - Connecticut Children's Medical Center - Hartford /ID# 137265, Hartford, Connecticut
  - Yale University School of Medicine /ID# 137257, New Haven, Connecticut
  - Nemours Children's Health System /ID# 148498, Jacksonville, Florida
  - University of Miami /ID# 140893, Miami, Florida
  - Winship Cancer Institute of Emory University /ID# 144274, Atlanta, Georgia
  - Children's Ctr Digestive, US /ID# 144625, Atlanta, Georgia
  - Children's Hospital New Orleans /ID# 144477, New Orleans, Louisiana
  - Maine Medical Partners /ID# 147685, Portland, Maine
  - Tufts Medical Center /ID# 143581, Boston, Massachusetts
  - Massachusetts General Hospital /ID# 141552, Boston, Massachusetts
  - Boston Children's Hospital /ID# 164102, Boston, Massachusetts
  - Duplicate_UMass Chan Medical School /ID# 148325, Worcester, Massachusetts
  - M Health Fairview University of Minnesota Medical Center - East Bank /ID# 137238, Minneapolis, Minnesota
  - Mayo Clinic - Rochester /ID# 149245, Rochester, Minnesota
  - Univ of Mississippi Med Ctr,US /ID# 137239, Jackson, Mississippi
  - Goryeb Children's Hospital /ID# 144275, Morristown, New Jersey
  - Women and Childrens Hosp /ID# 143778, Buffalo, New York
  - CCMC - Steven and Alexandra Cohen Children's Medical Center of New York /ID# 137266, New Hyde Park, New York
  - Columbia Univ Medical Center /ID# 144440, New York, New York
  - Columbia Univ Medical Center /ID# 144475, New York, New York
  - Univ Med Ctr at Stony Brook /ID# 140913, Stony Brook, New York
  - SUNY Upstate Medical University /ID# 148437, Syracuse, New York
  - Univ NC Chapel Hill /ID# 137236, Chapel Hill, North Carolina
  - Duke Cancer Center /ID# 137268, Durham, North Carolina
  - Children's Hospital Oklahoma /ID# 144047, Oklahoma City, Oklahoma
  - Geisinger Medical Center /ID# 149910, Danville, Pennsylvania
  - Penn State Child Hosp.Hersh,PA /ID# 144476, Hershey, Pennsylvania
  - Duplicate_Medical University of South Carolina /ID# 144473, Charleston, South Carolina
  - Children's Medical Center /ID# 149256, Dallas, Texas
  - Cook Children's Med. Center /ID# 144474, Fort Worth, Texas
  - Texas Children's Hospital /ID# 148211, Houston, Texas
  - University Of Vermont Medical /ID# 137263, Burlington, Vermont
  - Pediatric Specialty of VA /ID# 142831, Fairfax, Virginia
  - Duplicate_Swedish Medical Center /ID# 137258, Seattle, Washington
  - Seattle Children's Hospital /ID# 140879, Seattle, Washington
  - MultiCare Institute for Research & Innovation /ID# 152120, Tacoma, Washington
  - Children's Hospital Wisconsin - Milwaukee Campus /ID# 137259, Milwaukee, Wisconsin
- University Clinical Center Tuzla /ID# 130638, Tuzla, Tuzlanski, Bosnia and Herzegovina
- SHAT Hematologic Diseases /ID# 143572, Sofia, Bulgaria
- Canada (5):
  - Alberta Health Services /ID# 128717, Edmonton, Alberta
  - Duplicate_University of Manitoba / Health Scuience Centre / John Buhler Research /ID# 141310, Winnipeg, Manitoba
  - IWK Health Center /ID# 127912, Halifax, Nova Scotia
  - The Univ of Western Ontario /ID# 137962, London, Ontario
  - Hospital for Sick Children /ID# 127910, Toronto, Ontario
- Croatia (2):
  - Klinicki bolnicki centar Sestre milosrdnice /ID# 128256, Zagreb, City of Zagreb
  - Zadar General Hospital /ID# 129830, Zadar
- Czechia (5):
  - Fakultní nemocnice Hradec Králové - Sokolská /ID# 128521, Hradec Králové, Hradec Kralove
  - Fakultni Nemocnice Ostrava /ID# 127913, Ostrava, Ostrava-mesto
  - Fakultni nemocnice Olomouc /ID# 127437, Olomouc
  - Fakultni nemocnice Kralovske Vinohrady /ID# 127697, Prague
  - Krajska zdravotni a.s. Masarykova nemocnice v Usti nad Labem o.z. /ID# 129829, Ústí nad Labem
- Kobenhavns Universitet - Hvidovre Hospital (HH) /ID# 146013, Hvidovre, Capital Region, Denmark
- Estonia (2):
  - Tallinn Children's Hospital /ID# 126974, Tallinn, Harju
  - Children's Clinic Of Tartu Uni /ID# 146017, Tartu, Tartu
- France (2):
  - Duplicate_Hôpital Pierre Wertheimer /ID# 128193, Bron, Rhone
  - AP-HP - Hopital Necker /ID# 147702, Paris
- Germany (10):
  - Universitaetsklinikum Ulm /ID# 148444, Ulm, Baden-Wurttemberg
  - Duplicate_Universitaetsklinikum Erlangen /ID# 137274, Erlangen, Bavaria
  - Duplicate_Universitaetsklinikum Muenster /ID# 148441, Munster, Lower Saxony
  - Christliches Kinderhospital Osnabrueck /ID# 136629, Osnabrück, Lower Saxony
  - Universitaetsklinikum Aachen /ID# 126591, Aachen, North Rhine-Westphalia
  - Duplicate_Universitaetsklinikum Carl Gustav Carus an der TU Dresden /ID# 127696, Dresden, Saxony
  - Froehlich Gemeinschaftspraxis /ID# 127975, Forchheim
  - Duplicate_Universitaetsklinikum Freiburg /ID# 130010, Freiburg im Breisgau
  - Kinderarztpraxis Neuhausen /ID# 144402, Munich
  - Universitaetsklinikum Regensburg /ID# 137140, Regensburg
- Greece (5):
  - Agia Sofia Hospital /ID# 134349, Athens, Attica
  - General Hospital of Chest Diseases of Athens SOTIRIA /ID# 147690, Athens, Attica
  - Iatriko Kentro Athinon /ID# 130639, Marousi, Attica
  - Venizeleio General Hospital /ID# 147335, Heraklion
  - General Hospital of Thessaloniki Gennimatas /Id# 163658, Thessaloniki
- Our Lady's Hospital /ID# 127438, Manorhamilton, Leitrim, Ireland
- Israel (8):
  - Schneider Children's Medical Center /ID# 152683, Petah Tikva, Central District
  - Duplicate_Kaplan Medical Center /ID# 152945, Rehovot, Central District
  - Yitzhak Shamir Medical Center /ID# 157182, Ẕerifin, Central District
  - Shaare Zedek Medical Center /ID# 144277, Jerusalem, Jerusalem
  - Edmond And Lily Safra Children /ID# 148730, Ramat Gan, Tel Aviv
  - Duplicate_Ha'Emek Medical Center /ID# 156316, Afula
  - Rambam Health Care Campus /ID# 162061, Haifa
  - The Lady Davis Carmel Medical Center /ID# 151519, Haifa
- Italy (10):
  - ASST Fatebenefratelli Sacco - Ospedale Fatebenefratelli e Oftalmico /ID# 144279, Milan, Milano
  - Azienda Ospedaliero-Universitaria Policlinico Umberto I /ID# 141962, Rome, Roma
  - Ospedale Maggiore Carlo Alberto Pizzardi /ID# 147347, Bologna
  - Duplicate_A.O.U. Policlinico G. Martino /ID# 141683, Messina
  - ASST Fatebenefratelli Sacco/Ospedale dei Bambini Vittore Buzzi /ID# 141679, Milan
  - Duplicate_Universita di Napoli Federico II /ID# 144280, Naples
  - Duplicate_POLICLINICO PAOLO GIACCONE /ID# 138410, Palermo
  - Azienda Ospedaliera Ospedali Riuniti Villa Sofia Cervello /ID# 152684, Palermo
  - Azienda Ospedaliero-Universitaria di Parma /ID# 147441, Parma
  - Azienda Usl Di Pescara - Presidio Ospedaliero Di Pescara /ID# 141307, Pescara
- Lithuania (2):
  - Hospital of Lithuanian University of Health Sciences Kaunas Clinics /ID# 127809, Kaunas
  - Vilnius University Hospital Santaros Klinikos /ID# 127810, Vilnius
- Netherlands (2):
  - Duplicate_Academisch Medisch Centrum /ID# 141843, Amsterdam, North Holland
  - Duplicate_Erasmus Medisch Centrum /ID# 141841, Rotterdam, South Holland
- Portugal (2):
  - 2CA-Braga, Hospital de Braga /ID# 138269, Braga
  - Unidade Local de Saude Sao Joao, EPE /ID# 138146, Porto
- Puerto Rico (2):
  - Ctr. Gastroenterologia Ped Oes /ID# 140875, Mayagüez
  - San Jorge Children Hospital /ID# 138067, San Juan
- Romania (4):
  - Spitalul Clinic de Urgenta pentru Copii- Pediatrie II-Nefrologie Pediatrica /ID# 131297, Cluj-Napoca, Cluj
  - Spitalul Clinic de Urgenta pentru Copii ?Louis Turcanu? /ID# 130251, Timișoara, Timiș County
  - Spitalul Clinic de Urgenta Pentru Copii Grigore Alexandrescu /Id# 130358, Bucharest
  - Spitalul Clinic Judetean de Urgenta Targu Mures /ID# 137014, Târgu Mureş
- Spain (23):
  - Complejo Hospitalario Universitario A Coruña /ID# 137235, A Coruña, A Coruna
  - Hospital Arquitecto Marcide - Complejo Hospitalario Universitario de Ferrol /ID# 138462, Ferrol, A Coruna
  - Complejo Hospitalario Universitario de Santiago (CHUS) /ID# 141667, Santiago de Compostela, A Coruna
  - Hospital Universitari Son Espases /ID# 147446, Palma de Mallorca, Balearic Islands
  - Hospital Universitario Germans Trias i Pujol /ID# 139400, Badalona, Barcelona
  - Hospital Sant Joan de Deu /ID# 152059, Esplugues de Llobregat, Barcelona
  - Consorci Corporacio Sanitaria Parc Tauli Sabadell /ID# 149029, Sabadell, Barcelona
  - Hospital Universitario Severo Ochoa /ID# 141545, Leganés, Madrid
  - Hospital Universitario Puerta de Hierro - Majadahonda /ID# 157872, Majadahonda, Madrid
  - Hospital Clinico Universitario Virgen de la Arrixaca /ID# 138460, El Palmar, Murcia
  - Hospital Universitario Central de Asturias /ID# 163053, Oviedo, Principality of Asturias
  - OSI Ezkerraldea-Enkarterri-Cruces /ID# 141781, Barakaldo, Vizcaya
  - Hospital Universitario Vall d'Hebron /ID# 141778, Barcelona
  - Hospital Universitario Vall d'Hebron /ID# 146015, Barcelona
  - Hospital General de Granollers /ID# 140882, Barcelona
  - Hospital Universitario de Girona Doctor Josep Trueta /ID# 147572, Girona
  - Hospital Infantil Universitario Nino Jesus /ID# 165738, Madrid
  - Hospital Universitario 12 de Octubre /ID# 136998, Madrid
  - Hospital Universitario La Paz /ID# 161152, Madrid
  - Hospital Regional Universitario de Malaga /ID# 144289, Málaga
  - Compl Hospital Univer de Vigo /ID# 136999, Pontevedra
  - Hospital Universitario Dr. Peset /ID# 159484, Valencia
  - Hospital Universitario y Politecnico La Fe /ID# 141847, Valencia
- Sweden (2):
  - Karolinska University Hospital Solna /ID# 129045, Solna, Stockholm County
  - Sodersjukhuset /ID# 152685, Stockholm, Stockholm County
- United Kingdom (13):
  - University Hospital of Derby and Burton NHS Foundation Trust /ID# 131592, Derby, Derbyshire
  - Sheffield Children's Hospital NHS Foundation Trust /ID# 130370, Sheffield, England
  - Disc_Barts Health NHS Trust - The Royal London Hospital /ID# 128471, London, Greater London
  - University Hospital Southampton NHS Foundation Trust /ID# 147538, Southampton, Hampshire
  - Duplicate_NHS Greater Glasgow and Clyde /ID# 127436, Glasgow, Scotland
  - St Helier Hospital /ID# 150097, Carshalton, Surrey
  - NHS Grampian /ID# 131296, Aberdeen
  - Birmingham Women's and Children's NHS Foundation Trust /ID# 136631, Birmingham
  - Duplicate_Cambridge University Hospitals NHS Foundation Trust /ID# 143779, Cambridge
  - Alder Hey Children's Hospital /ID# 138013, Liverpool
  - Manchester University NHS Foundation Trust /ID# 128476, Manchester
  - Duplicate_The Newcastle Upon Tyne Hospitals NHS Foundation Trust /ID# 147438, Newcastle upon Tyne
  - St George's University Hospitals NHS Foundation Trust /ID# 131590, Tooting

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- See also: Related Info — http://www.rxabbvie.com